CLINICAL TRIAL: NCT04095858
Title: A Randomized, Double Blind, Placebo Controlled, Multi-center, Phase III Study of CD24Fc for Prevention of Acute Graft-Versus-Host Disease Following Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Efprezimod Alfa (CD24Fc, MK-7110) for the Prevention of Acute Graft Versus Host Disease (GVHD) Following Myeloablative Hematopoietic Stem Cell Transplantation (HSCT) (MK-7110-005)
Acronym: CATHY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Oncoimmune, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7110-005; 15-4789 (Other: FDA Orphan Drug Designation); FD-OOPD-006089 (Other Grant/Funding Number: FDA Orphan Products Clinical Trial Grant); CD24Fc-005 (Other: OncoImmune); MK-7110-005 (Other: Merck Protocol Number); NCT04976699 (obsolete NCT alias)
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Hematopoietic Stem Cell Transplantation; Acute Graft Versus Host Disease; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes | interventions — Sodium Chloride; Methotrexate; Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efprezimod alfa Treatment (Experimental): Efprezimod alfa: IV infusion, 480 mg (day -1), 240 mg (day +14) and 240 mg (day +28); Tacrolimus: begin on day -3. IV [0.03 mg/kg/day] or by mouth (PO) [0.045 mg/kg/dose] dosing is permitted; Methotrexate: given IV at a dose of 15 mg/m^2/dose once daily on Day 1 after hematopoietic cell transplantation (HCT), and at a dose of 10 mg/m^2/dose on days 3, 6, and 11 after HCT.
  Interventions: Drug: Efprezimod alfa; Drug: Methotrexate; Drug: Tacrolimus
- Placebo (Placebo Comparator): Placebo (Saline solution): 100 ml IV infusion, Day -1, Day 14, Day 28. Tacrolimus: begin on day -3. IV [0.03mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted; Methotrexate: given IV at a dose of 15 mg/m^2/dose once daily on Day 1 after HCT, and at a dose of 10 mg/m^2/dose on days 3, 6, and 11 after HCT.
  Interventions: Drug: Placebo; Drug: Methotrexate; Drug: Tacrolimus

INTERVENTIONS:
Drug: Efprezimod alfa — IV infusion: 480 mg at Day -1, 240 mg at Day 14, 240 mg at Day 28.
  Other Names: Human CD24 and human IgG Fc Fusion Protein; MK-7110
  Arms: Efprezimod alfa Treatment
Drug: Placebo — IV infusion, 100 ml at Day -1, Day 14, and Day 28.
  Other Names: Saline
  Arms: Placebo
Drug: Methotrexate — IV, 15 mg/m^2/dose at Day 1, then 10 mg/m2/dose at Day 3, 6, 11.
  Other Names: Trexall
Drug: Tacrolimus — Begin on day -3. IV [0.03 mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted
  Other Names: FK506; Prograf

SUMMARY:
The study compares two acute graft-versus-host disease (aGVHD) prophylaxis regimens: efprezimod alfa vs placebo with the standard GVHD prophylaxis of tacrolimus / methotrexate.

The study compares two acute graft-versus-host disease (aGVHD) prophylaxis regimens: efprezimod alfa/tacrolimus / methotrexate (efprezimod alfa/Tac/MTX) versus placebo/tacrolimus / methotrexate (placebo/Tac/MTX) in the setting of myeloablative conditioning (MAC), matched unrelated donor (MUD) allogeneic hematopoietic stem cell transplantation in participants with acute leukemia (AML/ALL) or myelodysplastic syndrome (MDS). The study agent, efprezimod alfa, will be administered through IV infusion on days -1, 14, and 28 at the dose of 480mg, 240 mg and 240mg, respectively. The placebo will be 100 ml normal saline intravenous (IV) solution.

DETAILED DESCRIPTION:
The Sponsor decided to discontinue screening and enrollment in this study on 18 May 2021 for business reasons. This decision was not related to any new or unexpected safety or efficacy findings.

ELIGIBILITY:
Inclusion Criteria:

1. A prospective participant for allogeneic HCT for a malignant hematologic disorder.
2. The donor and recipient must have a human leukocyte antigen (HLA)-8/8 allelic match at the HLA-A, -B, -C, and - DRB1 loci. High-resolution typing is required for all alleles for unmatched donors. Only matched unrelated donors are acceptable for this trial.
3. The following diagnoses are to be included:

   1. Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL) in first or second remission. Remission is defined as the absence of blasts in the peripheral circulation at the time of enrollment, < 5% blasts in the bone marrow and absence of extramedullary disease including CNS involvement.
   2. Myelodysplastic syndrome (MDS) with intermediate or high-risk International Prognostic Scoring System (IPSS) or equivalent Revised International Prognostic Scoring System (IPSS-R) score with < 10% blasts in the bone marrow.
4. Males or non-pregnant, non-lactating females, ≥ 18 years of age. Note there is no defined upper age limited, so long as deemed appropriate candidate for myeloablative conditioning.
5. Karnofsky Performance Status >70%.
6. Participants must have normal or near normal organ function as defined by their treating institutions bone marrow transplant (BMT) program clinical practice guidelines. In addition, for purposes of this protocol minimum organ function criteria within 30 days of beginning conditioning include: Eligibility According to Pre HCT Organ Function:

   1. Total bilirubin ≤2.5 mg% (unless from Gilbert's disease or disease-related);
   2. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT))/ alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SGPT)) <5.0 X institutional upper limit of normal;
   3. Estimated or actual glomerular filtration rate (GFR)>50 mL/min/1.73 m2 for participants with creatinine levels above institutional normal (GFR should be corrected for BSA);
   4. Pulmonary Function Tests include diffusing capacity of the lungs for carbon monoxide (DLCO), forced expiratory volume in one second (FEV1), forced vital capacity (FVC)> 50% DLCO should be corrected for hemoglobin;
   5. Ejection Fraction >50%;
   6. Hematopoietic Cell Transplantation-Specific Comorbidity Index (HCT-CI) ≤ 5.

   Item d and e may be assessed up to 10 weeks prior to the start of conditioning therapy.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Women of child bearing potential and men must agree to use contraception prior to study entry and through day 100 post HCT (hormonal or barrier method of birth control; abstinence). Should a woman become pregnant or suspect she is pregnant while she or her partner is on treatment in this study, she should inform her study physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study until day 100 post HCT.

Exclusion Criteria:

1. Subjects may not have presence of active central nervous system (CNS) disease or extramedullary disease.
2. Prior cytotoxic chemotherapy within 21 days from the initiation of HCT conditioning (i.e. intensive induction / consolidation for AML). Note, certain low intensity treatments not intended to induce remission but rather stabilize disease are acceptable up to 24 hrs prior to initiation of HCT conditioning (i.e. Tyrosine Kinase Inhibitor, sorafenib).
3. Cord blood and haploidentical donors are not eligible.
4. HLA-mismatch at the HLA-A, -B, -C, and - DRB1 loci. Note, HLA-DQ mismatches are permissible.
5. Pregnant and nursing mothers are excluded from this study. This is because the risk to the fetus is unknown.
6. Any physical or psychological condition that, in the opinion of the investigator, would pose unacceptable risk to the participant or raise concern that the participant would not comply with protocol procedures.
7. Uncontrolled infections. Participants still under therapy for presumed or proven infection are eligible provided there is clear evidence (radiologic, clinical and/or culture) that the infection is well controlled.
8. Participants seropositive or polymerase chain reaction (PCR) positive for the human immunodeficiency virus (HIV). Participants with evidence of Hepatitis B or Hepatitis C PCR positivity.
9. Prior HCT (allograft or prior autograft).
10. Use of T cell depletion either ex vivo or in vivo (i.e. anti-thymocyte globulin (ATG), alemtuzumab) is prohibited.
11. Current or prior diagnosis of antecedent Myelofibrosis is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - City of Hope ( Site 0302), Duarte, California
  - The University of Chicago Medical Center ( Site 0306), Chicago, Illinois
  - Penn State University Milton S. Hershey Medical Center ( Site 0304), Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania ( Site 0309), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 6 sites in the United States.
Pre-assignment Details: Eleven participants were screened but the decision was made to terminate the study after only 7 were randomized and treated in one of the study arms.
Groups:
- Placebo Treatment: Placebo (Saline solution): 100 ml IV infusion, Day -1, Day 14, Day 28. Tacrolimus: begin on day -3. IV [0.03mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted; Methotrexate: given IV at a dose of 15 mg/m^2/dose once daily on Day 1 after HCT, and at a dose of 10 mg/m^2/dose on days 3, 6, and 11 after HCT.
- CD24Fc Treatment: CD24Fc: IV infusion, 480 mg (day -1), 240 mg (day +14) and 240 mg (day +28); Tacrolimus: begin on day -3. IV [0.03 mg/kg/day] or by mouth (PO) [0.045 mg/kg/dose] dosing is permitted; Methotrexate: given IV at a dose of 15 mg/m^2/dose once daily on Day 1 after hematopoietic cell transplantation (HCT), and at a dose of 10 mg/m^2/dose on days 3, 6, and 11 after HCT.
Period: Overall Study
Arm/Group | Placebo Treatment | CD24Fc Treatment
Started | 3 | 4
Completed | 0 | 0
Not Completed | 3 | 4
Not completed — Death | 1 | 0
Not completed — Study terminated by Sponsor | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CD24Fc Treatment | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (16.46) | 45.0 (8.29) | 38.6 (13.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 180 Day Grade III-IV Acute Graft-Versus-Host Disease (GVHD)-Free Survival (aGFS)
Description: Grade III-IV aGFS was defined as the time in days to the earlier of the first documented acute Grade III-IV GVHD or death by any cause in 180 days after hematopoietic stem cell transplantation (HCT). Event grading was based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 criteria. Participants who did not drop out or experience aGVHD or death were censored at the time of leukemia relapse or Day 180, whichever came first.
Time Frame: Up to 180 days after HCT
Population: All randomized participants are included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | CD24Fc Treatment
Number analyzed (Participants) | 3 | 4
days | NA [45.0 to NA] — Median and upper limit of 95% CI not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — Median (95% CI) not reached at time of data cut-off due to insufficient number of participants with an event.

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from HCT to death due to any cause. Participants who were alive at the end of the 180 days post HCT were censored at the last date they were known to be alive.
Time Frame: Up to 180 days after HCT
Population: All randomized participants are included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | CD24Fc Treatment
Number analyzed (Participants) | 3 | 4
days | NA [45.0 to NA] — Median and upper limit of 95% CI not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — Median (95% CI) not reached at time of data cut-off due to insufficient number of participants with an event.

3. Secondary Outcome: Disease Free Survival (DFS)
Description: DFS is defined as the earlier of time to leukemia relapse, or death, whichever occurred first. Subjects that were alive and did not experience disease relapse at the end of the follow-up period (180 days after HCT) were censored at the last date of evaluation.
Time Frame: Up to 180 days after HCT
Population: All randomized participants are included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | CD24Fc Treatment
Number analyzed (Participants) | 3 | 4
days | NA [45.0 to NA] — Median and upper limit of 95% CI not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — Median (95% CI) not reached at time of data cut-off due to insufficient number of participants with an event.

4. Secondary Outcome: 180 Day Grade II-IV aGFS
Description: Grade II-IV aGFS was defined as the time in days to the earlier of the first documented acute Grade II-IV GVHD or death by any cause in 180 days after HCT. Event grading was based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 criteria. Participants who did not drop out or experience aGVHD or death were censored at the time of leukemia relapse or Day 180, whichever came first.
Time Frame: Up to 180 days after HCT
Population: All randomized participants are included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | CD24Fc Treatment
Number analyzed (Participants) | 3 | 4
days | 45.0 [29.0 to 56.0] | NA [28.0 to NA] — Median and upper limit of 95% CI not reached at time of data cut-off due to insufficient number of participants with an event.

5. Secondary Outcome: 180 Day Grade III-IV aGVHD-free and Relapse-free Survival (aGVHD RFS)
Description: Grade III-IV aGVHD RFS was defined as the time in days to the earlier of the first documented acute Grade III-IV aGVHD, relapse, or death by any cause in 180 days after HCT. Event grading was based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 criteria. Participants who did not drop out, experience Grade III-IV aGVHD, relapse, or death were censored at Day 180.
Time Frame: Up to 180 days after HCT
Population: All randomized participants are included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | CD24Fc Treatment
Number analyzed (Participants) | 3 | 4
days | NA [45.0 to NA] — Median and upper limit of 95% CI not reached at time of data cut-off due to insufficient number of participants with an event. | NA [28.0 to NA] — Median (95% CI) not reached at time of data cut-off due to insufficient number of participants with an event.

ADVERSE EVENTS:
Time Frame: Up to 180 days
Description: All participants who received ≥1 dose of study therapy are included in assessment of adverse events (AEs) and serious AEs (SAEs). All-cause mortality was assessed in all randomized participants.
Arm/Group | Placebo | CD24Fc Treatment
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | CD24Fc Treatment (N=4)
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | CD24Fc Treatment (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Chronic graft versus host disease oral (Immune system disorders) | 0 | 1
Graft versus host disease in skin (Immune system disorders) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Vascular access site discharge (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site erythema (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Claustrophobia (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Blue toe syndrome (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Platelet count decreased (Investigations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT04095858/Prot_SAP_000.pdf